CLINICAL TRIAL: NCT04697238
Title: Effect of Artificial Loading, Through Application of Weight Vests, on Body Weight in Obese Subjects; a Randomized Controlled Trial
Brief Title: Anti-obesity Treatment by Loading in Adult Subjects
Acronym: ATLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATLAS
Record Dates: First submitted 2020-12-14; First posted 2021-01-06 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: A parallel study design will be used in which the control group is to be compared with the intervention group. To avoid the risk of carry-over effects, the investigators have decided to not use a crossover design. This could have decreased the variation of the measurement values and increased the power of the study. However, the investigators believe there could be a risk of a carry-over effect with a cross over design. As this is a new effect in clinical studies, the investigators have no information about the wash-out time needed to avoid this problem.
Who Masked: Outcomes Assessor
Masking Description: Subjects might be able to determine if they are in the control group or intervention group since it is difficult to mask the difference between a heavy and a light weight vest. Therefore, intervention in this study won't be masked for the participants. However, group affiliation will be masked for outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High load (11 % of body weight vests) (Experimental): Subjects in this arm will carry heavy weight (11 percent of body weight) vests for 5 weeks.
  Interventions: Device: Weight vest
- Low load (1 % of body weight vests) (Placebo Comparator): Subjects in this arm will carry heavy weight (1 percent of body weight) vests for 5 weeks.
  Interventions: Device: Weight vest

INTERVENTIONS:
Device: Weight vest — A vest weighing up to a maximum of 15 kg.
  Other Names: Artificial weights

SUMMARY:
Obesity related ailments, such as cardiovascular diseases (CVD) and metabolic disorders are major causes of death in the Western World. This trial may result in improved prevention, diagnosis and treatments for obesity and obesity-related disorders. Published data show that if a weight is carried by a rodent, this animal will lose body weight and gain an improved glucose control. Recently published data further show comparable results in humans when carrying an additional weight.

The investigators aim to confirm and further investigate these findings in humans. The investigators plan to let obese participants carry weight vests and monitor their change in body weight. The investigators will also measure food intake, physical activity, energy expenditure, body composition, abdominal fat and heart rate variability. This to further examine the potential beneficial effects of loading and the mechanism of action.

DETAILED DESCRIPTION:
STUDY OBJECTIVES AND ENDPOINTS

Primary objective

To determine if wearing a weight vest with 11 percent of body weight for 8 hours/day for 5 weeks decreases body weight in obese subjects.

Secondary objectives

To determine if wearing a weight vest with 11 percent of an individual's body weight for up to 5 weeks affects levels of abdominal fat, liver fat, fat mass, fat free mass, physical activity, energy expenditure, waist circumference, food intake or activity in the autonomic nervous system in obese subjects.

To determine, exploratory, if wearing a weight vest with 11 percent of an individual's body weight for up to 5 weeks affects serum concentrations of circulating proteins, metabolites or electrolytes in obese subjects.

STUDY DESIGN AND PROCEDURES

Overall study design and procedure protocol

The aim of the study is to investigate the effect of adding artificial weights to individuals suffering from obesity. Enrolled study subjects will be randomized in a 1:1 fashion to either carry a heavy weight vest with 11 percent of the individual's body weight (intervention group) or a light weight vest with 1 percent of the individual's body weight (control group). The weight vests will be worn for a total of 5 weeks.

Body weight, abdominal fat, liver fat, waist circumference, food intake, energy expenditure, physical activity, activity in the autonomic nervous system, fat mass, bone mass, water mass and fat free mass together with endpoint blood samples will be measured before the start of intervention to obtain base line values. New measurements will then be done for comparison during or after the intervention to determine the effect of added artificial loading on obese subject.

The study consists of a total of 10 weeks. During the first 3 weeks of the study measurements will be made which will be used as baseline. The following 5 weeks contains the intervention and the carrying of a weight vest. The last 2 weeks is a follow up period and at the end of this period follow up measurements will be done. During or after the intervention period new measurements will be made to be compared with the baseline measurements to evaluate the study endpoints.

To avoid the risk of carry-over effects, the investigators have decided to not use a crossover design. This could have decreased the variation of the measurement values and increased the power of the study. However, the investigators believe there could be a risk of a carry-over effect with a cross over design. As this is a completely new effect in clinical studies, the investigators have no information about the wash-out time needed to avoid this problem.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Consent out of free will.
3. 18-65 years of age.
4. Obesity as defined by a BMI >30 and ≤35. Fat mass > 25 %.
5. Willingness to comply with the study protocol
6. Normal or clinically non-significant screening of blood samples:

   1. Hemoglobin (Hb), White Blood Cell Count (WBC), thrombocyte count, sodium (Na), potassium (K), chloride (Cl), calcium (Ca), creatinine, aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), total bilirubin, Prothrombin Time (PT-INR), Activated Partial Thromboplastin Time (APTT), human immunodeficiency viruses (HIV), Hepatitis B, Hepatitis C, glycated hemoglobin (HbA1c), C-reactive protein (CRP), free thyroxine (fT4), thyroid-stimulating hormone (TSH).
   2. Normal or clinically non-significant aberrations of screening blood samples are defined as:

   i. Normal: Values within the reference interval supplied by the local lab at Sahlgrenska University Hospital

   ii. Clinically non-significant aberration: as judged by investigator (Clinical significance judged by investigator)
7. Normal or non-clinically significant 12-lead electrocardiography (ECG) recording as judged by the investigator.

Exclusion Criteria:

1. Chronic disease that could interfere with the participation in the study as judged by the investigator. For example poorly regulated type 1 or 2 diabetes, severe cardiovascular disease that effect daily life, severe pulmonary disease that affects daily life or malignancy.
2. Chronic pain such as pain that is constant and impairs quality of life as judged by the investigator; for example: significant back, hip and knee pain.
3. Regular consumption of medicine or natural supplements that affect weight, inhibit physical activity or increase the risk of adverse effects as judged by the investigator. The following drugs will not be accepted:

   1. β-blockers, Glucagon-like peptide-1 (GLP-1) agonists, Dipeptidyl peptidase-4 (DPP-IV) inhibitors, SGLT2-inhibitors, sulfonylureas, insulin, orlistat, anti-obesity drugs, antidepressants, bisphosphonates, β2-agonists, oral corticosteroids, diuretics, benzodiazepines, or central nervous system stimulating drugs such as methylphenidate or dextroamphetamine.
   2. Any illegal drugs according to local laws and regulation
4. Gastric by-pass surgery or equivalent metabolic surgery in the gastrointestinal tract.
5. Reduced mobility.
6. Pregnancy. Females of childbearing potential must confirm to use reliable contraception (intrauterine device, oral contraceptives or condom) and not suspect to be pregnant. Pregnancy test will be taken on all female subjects of fertile age unless permanently sterile, as judged by the investigator. Permanently sterile women can be excluded from the pregnancy test. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy
7. Change in body weight of 5 kg or greater during the past 3 months or recently started a strict diet. Also, a greater change in body weight than 4 kg difference between day -21 and day 0 will not be accepted.
8. Use of any illegal drugs according to local regulations or consuming excessive amounts of alcohol, tobacco, nicotine.

   a. Excessive amounts of above-mentioned substances defined as:

   i. Consumption of more than 9 glasses of wine for women, 14 glasses of wine for men (15 cl/glass 11 % alcohol) or equivalent as judged by investigator during an ordinary week will not be accepted.

   ii. Individuals with a consumption equal or higher than 10 cigarettes or half a packet of snuff per day.
9. Drastic change in lifestyle during the last 3 months; for example a significant change in physical activity, dietary habits, nicotine, alcohol or drug use as judged by the investigator.
10. Apparent risk of not being able to comply with the study protocol for any reason as judged by the investigator.
11. Having participated in a similar study during the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Change in body weight at 5 weeks | 35 days
  Change in body weight (in percent of baseline body weight) between day 35 and baseline in the high load group compared with low load group.

SECONDARY OUTCOMES:
Change in body weight at 15 days | 15 days
  Change in body weight between day 15 and baseline measured in grams.
Change in subcutaneous fat at 35 days | 35 days
  Change in levels of subcutaneous fat between day 35 and baseline measured in cm^2 from CT images of the abdomen.
Change in visceral fat at 35 days | 35 days
  Change in levels of visceral fat between day 35 and baseline measured in cm^2 from CT images of the abdomen.
Change in liver fat at 35 days | 35 days
  Change in levels of liver fat between day 35 and baseline measured in Hounsfield Units (HU) from CT images of the abdomen.
Change in body composition at 35 days | 35 days
  Change in levels of fat mass and fat free mass between day 35 and baseline measured in grams with Dual-energy X-ray absorptiometry (DXA).
Change in waist circumference at 35 days | 35 days
  Change in waist circumference between day 35 and baseline measured in centimeters with measuring tape.
Change in physical activity at 21 days | 21 days
  Change in physical activity between day 21 and baseline. Measured as time distribution in a spectrum of physical activity intensities assessed by accelerometer worn for 24 hours a day for one week. Change measured in minutes per day. Changes compared between measurements during intervention (day 15 to 21) and baseline (day -13 to -7).
Change in energy expenditure at 28 days | 28 days
  Change in energy expenditure between day 28 and baseline measured in joules per day with the doubly labeled water method. Changes compared between measurement during intervention (day 14 to 28) and baseline (day -14 to 0).
Change in food intake at 28 days | 28 days
  Change in food intake between day 28 and baseline measured in calories with the validated questionnaire Short Dietary Questionnaire (SDQ). Changes compared between measurement during intervention (day 14 to 28) and baseline (day -14 to 0).
Change in autonomic nervous system activity at 15 days | 15 days
  Change in heart rate variability (HRV) between day 15 and baseline measured in milliseconds with 24-hour electrocardiography (ECG) monitoring. Changes measured at day 15 compared with baseline (day -13).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Curiac, Principal Investigator — Clinical Trial Center, Sahlgrenska University Hospital
Locations (1):
- Clinical Trial Center, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jansson JO, Palsdottir V, Hagg DA, Schele E, Dickson SL, Anesten F, Bake T, Montelius M, Bellman J, Johansson ME, Cone RD, Drucker DJ, Wu J, Aleksic B, Tornqvist AE, Sjogren K, Gustafsson JA, Windahl SH, Ohlsson C. Body weight homeostat that regulates fat mass independently of leptin in rats and mice. Proc Natl Acad Sci U S A. 2018 Jan 9;115(2):427-432. doi: 10.1073/pnas.1715687114. Epub 2017 Dec 26. PMID 29279372
- [Background] Ohlsson C, Gidestrand E, Bellman J, Larsson C, Palsdottir V, Hagg D, Jansson PA, Jansson JO. Increased weight loading reduces body weight and body fat in obese subjects - A proof of concept randomized clinical trial. EClinicalMedicine. 2020 Apr 30;22:100338. doi: 10.1016/j.eclinm.2020.100338. eCollection 2020 May. PMID 32510046
- [Derived] Bellman J, Westerterp K, Wouters L, Johannesson M, Lundqvist N, Kullberg J, Larsson C, Gustafsson M, Pettersson S, Fridolfsson J, Arvidsson D, Borjesson M, Curiac D, Jansson JO, Jansson PA, Ohlsson C. Increased weight-load improves body composition by reducing fat mass and waist circumference, and by increasing lean mass in participants with obesity: a single-centre randomised controlled trial. BMC Med. 2025 May 30;23(1):317. doi: 10.1186/s12916-025-04143-6. PMID 40442671